CLINICAL TRIAL: NCT06476977
Title: Trigger Finger Corticosteroid Injection Pain: Palmar Injection Versus Dorsal Intrasynovial (Transthecal) Injection
Brief Title: Intrasynovial Digital Anesthesia in Trigger Finger
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kevin Zuo (Other)
Responsible Party: Sponsor-Investigator, Kevin Zuo, Staff Surgeon, Plastic and Reconstructive Surgery, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-5288
Record Dates: First submitted 2024-06-20; First posted 2024-06-27 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Trigger Finger Disorder
Keywords: trigger finger; stenosing tenosynovitis; corticosteroid injection; palmar; dorsal; pain
MeSH Terms: conditions — Trigger Finger Disorder; Tendon Entrapment; Pain | interventions — Anesthetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dorsal Webspace Approach (Experimental): A dorsal approach involves passing the needle with a 1:1 triamcinolone and lidocaine mixture in the dorsal webspace skin aiming just palmar to the proximal phalanx bone such that the needle is directed into the flexor tendon sheath at the A1 annular pulley.
  Interventions: Procedure: Dorsal webspace combined corticosteroid and anesthetic injection
- Palmar Approach (Active Comparator): Standard approach for injecting the 1:1 triamcinolone and lidocaine mixture involves the needle passing through the cutaneous and subcutaneous layers of the palmar skin surface and into the flexor tendon sheath at the A1 annular pulley.
  Interventions: Procedure: Palmar combined corticosteroid and anesthetic injection

INTERVENTIONS:
Procedure: Dorsal webspace combined corticosteroid and anesthetic injection — The dorsal webspace injection consists of a 1cc mixture of 0.5cc triamcinolone (Kenalog) 10mg/mL and 0.5cc 1% lidocaine for analgesic purposes.
  Arms: Dorsal Webspace Approach
Procedure: Palmar combined corticosteroid and anesthetic injection — The palmar injection consists of a 1cc mixture of 0.5cc triamcinolone (Kenalog) 10mg/mL and 0.5cc 1% lidocaine for analgesic purposes.
  Arms: Palmar Approach

SUMMARY:
Trigger finger is a common disease of the hand involving swelling and inflammation of the tendon which flexes a finger, causing catching, locking, and/or pain. Trigger finger is typically treated by hand surgeons with a steroid injection through the front/palm side of the hand into the area near the tendon (i.e., at the base of the affected finger). This steroid injection is often combined with a local anesthetic (numbing agent) to help reduce short-term pain from the injection. However, the front/palm side of the hand is known to be very sensitive, and the steroid injection can be quite painful as the needle pierces the front/palm skin.

To reduce the pain of steroid injections for trigger finger, a different approach involves performing the injection from the back/dorsal side of the hand, which is thought to be less sensitive (and therefore less painful) than the front/palm side of the hand. This technique is sometimes used and has been previously studied, but it is not clear if it can offer less injection-related pain than standard treatment.

Accordingly, this study will be comparing short-term injection-associated pain between front/palm side and back/dorsal side steroid injections for trigger finger. The study will also seek to understand what area of the hand is numbed by the anesthetic when doing a front/palm side injection versus a back/dorsal side injection of the hand. Overall, the investigators hypothesize that back/dorsal side injections will be less painful than front/palm side injections for trigger fingers and that the area of numbing from the anesthetic will be equivalent between both types of injections.

DETAILED DESCRIPTION:
Trigger finger (stenosing tenosynovitis) is one of the most common pathologies assessed by hand surgeons in clinic. Trigger finger involves inflammation or edema of the flexor tendon causing friction of the tendon at the site of the A1 annular pulley located at the base of the affected finger in the palm. Trigger finger is typically managed non-surgically in a clinic setting with percutaneous corticosteroid injection (CSI) which can be successful in alleviating symptoms. Patients with trigger finger who do not respond to CSI, have incomplete relief, and/or who have recurrent symptoms may then receive surgical management with release of the A1 pulley.

CSIs for trigger fingers are among the most common procedures performed by hand surgeons and are often administered multiple times in a single clinic day. CSIs are frequently mixed 50:50 with 1% lidocaine to provide post-injection analgesia for patients as well as symptomatic relief of the trigger finger if acutely inflamed. These injections are commonly administered from a palmar approach into the A1 pulley of the affected digit. Numerous technical variations of palmar trigger finger injections have been described involving either subcutaneous injection superficial to the flexor tendon sheath or intrasynovial (transthecal) injection into the flexor tendon sheath.

Unfortunately, given the rich sensory innervation of the palmar skin, palmar injections are associated with significant pain as the needle pierces the skin. An alternative technique is to provide digital anesthesia from a dorsal webspace approach, injecting the local anesthetic into the flexor tendon synovial sheath. This intrasynovial or transthecal technique has the benefit of a dorsal approach where the skin is less sensitive resulting in less pain (6). This technique has been described previously but is not familiar to many hand surgeons and is not routinely used in North America.

Anecdotally, patients report significantly decreased pain with the dorsal intrasynovial injection technique for trigger finger injections, but pain scores have not been quantitatively evaluated or compared to the pain scores of traditional palmar trigger finger injections. Furthermore, it is not known what distribution of digital sensory blockade is achieved with this intrasynovial technique, particularly on the dorsal surface of the digit which is discontinuous with the flexor tendon sheath and innervated by the sensory branch of the radial nerve.

Accordingly, it is hypothesized that injecting corticosteroids into the synovial sheath of the flexor tendon will result in less pain over 24 hours if performed through the dorsal webspace versus the palmar side of the affected digit.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older
* Have a diagnosis of trigger finger (can be any of the 5 digits)
* Opting to receive a CSI for their triggering finger

Exclusion Criteria:

* Decline to obtain a CSI for trigger finger management
* Receiving multiple CSI for trigger finger management at the appointment
* Past CSI and/or surgery to the digit involved
* Unable to communicate in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) - Pain | measured at 0 hours, 4 hours, and 24 hours post-injection
  100mm mechanical rating scale for pain, ranging from 0mm ("no pain") to 100mm ("pain as bad as it could be"); higher scores indicate a worse outcome.
Numerical Rating Scale (NRS) - Pain | measured at 0 hours, 4 hours, and 24 hours post-injection
  11-point numerical rating scale for pain, ranging from 0 (no pain) to 10 (worst pain ever possible); higher scores indicate a worse outcome.
Short-Form McGill Pain Questionnaire (SFMPQ) - Present Pain Intensity (PPI) | measured at 0 hours, 4 hours, and 24 hours post-injection
  5-point combined numerical-word rating scale for pain, ranging from 1 (mild) to 5 (excruciating); higher scores indicate a worse outcome.

SECONDARY OUTCOMES:
Sensory Assessment - Light Touch | measured at 0 hours post-injection
  Semmes-Weinstein 2.0g monofilament test as threshold of sensory impairment
Sensory Assessment - Pain | measured at 0 hours post-injection
  Pinprick pain sensation with an 18-gauge sharp needle tip

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Zuo, MD, MASc, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network - Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Akhtar S, Bradley MJ, Quinton DN, Burke FD. Management and referral for trigger finger/thumb. BMJ. 2005 Jul 2;331(7507):30-3. doi: 10.1136/bmj.331.7507.30. No abstract available. PMID 15994689
- [Background] Makkouk AH, Oetgen ME, Swigart CR, Dodds SD. Trigger finger: etiology, evaluation, and treatment. Curr Rev Musculoskelet Med. 2008 Jun;1(2):92-6. doi: 10.1007/s12178-007-9012-1. PMID 19468879
- [Background] Fleisch SB, Spindler KP, Lee DH. Corticosteroid injections in the treatment of trigger finger: a level I and II systematic review. J Am Acad Orthop Surg. 2007 Mar;15(3):166-71. doi: 10.5435/00124635-200703000-00006. PMID 17341673
- [Background] Merry SP, O'Grady JS, Boswell CL. Trigger Finger? Just Shoot! J Prim Care Community Health. 2020 Jan-Dec;11:2150132720943345. doi: 10.1177/2150132720943345. PMID 32686570
- [Background] Patrinely JR Jr, Johnson SP, Drolet BC. Trigger Finger Corticosteroid Injection With and Without Local Anesthetic: A Randomized, Double-Blind Controlled Trial. Hand (N Y). 2021 Sep;16(5):619-623. doi: 10.1177/1558944719884663. Epub 2019 Nov 5. PMID 31690121
- [Background] Jimenez I, Garces GL, Marcos-Garcia A, Medina J. A randomized controlled trial of dorsal web space versus palmar midline injection of steroid in the treatment of trigger digits. J Hand Surg Eur Vol. 2020 Dec;45(10):1071-1077. doi: 10.1177/1753193420927999. Epub 2020 Jun 3. PMID 32493111
- [Background] Bitar H, Zachrisson AK, Bystrom M, Stromberg J. Day-by-day symptom relief after corticosteroid injection for trigger digit: a randomized controlled study of two techniques. J Hand Surg Eur Vol. 2023 Oct;48(9):849-856. doi: 10.1177/17531934231177422. Epub 2023 May 22. PMID 37218106
- [Background] Rosenbaum YA, Benvenuti N, Yang J, Ruff ME, Awan HM, Samora JB. The Effect of Trigger Finger Injection Site on Injection-Related Pain. Hand (N Y). 2018 Mar;13(2):164-169. doi: 10.1177/1558944717703134. Epub 2017 Apr 26. PMID 28443675
- [Background] Mathew A. Mid-axial injection of steroid into the flexor sheath for trigger fingers. J Hand Microsurg. 2014 Jun;6(1):49-52. doi: 10.1007/s12593-014-0120-z. Epub 2014 Feb 21. No abstract available. PMID 24876694
- [Background] Jimenez I, Medina J, Marcos-Garcia A, Garces GL. Out-of-sheath corticosteroid injections through the dorsal webspace for trigger finger and trigger thumb. A prospective cohort study. Rev Esp Cir Ortop Traumatol. 2022 Jul-Aug;66(4):260-266. doi: 10.1016/j.recot.2021.03.009. Epub 2021 Aug 6. English, Spanish. PMID 34366261
- [Background] Haefeli M, Elfering A. Pain assessment. Eur Spine J. 2006 Jan;15 Suppl 1(Suppl 1):S17-24. doi: 10.1007/s00586-005-1044-x. Epub 2005 Dec 1. PMID 16320034
- [Background] Melzack R. The McGill Pain Questionnaire: major properties and scoring methods. Pain. 1975 Sep;1(3):277-299. doi: 10.1016/0304-3959(75)90044-5. PMID 1235985